CLINICAL TRIAL: NCT06568575
Title: The Effects of Exercise and Music Combination on Sports Anxiety, Exercise Beliefs, Coping Effectiveness, and Mental Toughness Among Chinese Sports Anxiety College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Liu Zhutang, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23040346
Record Dates: First submitted 2024-08-14; First posted 2024-08-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Health; Sports Anxiety; Mental Toughness; Coping Effectiveness; Exercise Beliefs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group of combine of exercise and music (Experimental): This study held a group meeting before the formal experiment to guide all participants in advance and describe the entire experimental process in detail to them. Students who had questions were given a unified and detailed explanation. Each participant received an instruction manual and a sports smart bracelet. During the experimental stage, the researcher would remind the participants on time to conduct the music and jogging experiment. The participants were required to participate in the experiment according to the contents of the instruction manual and upload each experimental participation content in the form of video or photos to the online information collection link posted by the participants. before experiment, 4 weeks, 8 weeks and 12 weeks，this study required participants to fill out the questionnaire four times.
  Interventions: Behavioral: experiment of music; Behavioral: experiment of exercise
- Control group (No Intervention): At the same time as the experimental group, a booklet about music and exercise was distributed to the participants. The control group and the experimental group had the same time to fill in the questionnaire. The control group was asked to fill in the first questionnaire before the experiment. After 4 weeks, the control group was asked to fill in the second questionnaire. After 8 weeks, the control group was asked to fill in the third questionnaire. After 12 weeks, the control group was asked to fill in the fourth questionnaire。After the study completed, the control group was also provided with the music and jogging materials for their reference. So that they received the same benefit as the experimental group.

INTERVENTIONS:
Behavioral: experiment of music — Participants in this study were randomly divided into a control group and an experimental group. The control group did not intervene, and they continued their normal routine. Participants in the control group were asked not to participate in additional physical activity or sports during the study period. The experimental group was intervened by exercise program. During the experimental experiment phase, all participants were asked to be in similar environments as possible: sports environment, living environment, and disturbed environment. The exercise experiment was 3 times a week with a period of 12 weeks. The length of time was 40 minutes each time and a total experiment time of 1420 minutes.
  Arms: experimental group of combine of exercise and music
Behavioral: experiment of exercise — Participants in this study were randomly divided into a control group and an experimental group. The control group did not intervene, and they continued their normal routine. Participants in the control group were asked not to participate in additional physical activity or sports during the study period. The experimental group was intervened by music program. During the experimental experiment phase, all participants were asked to be in similar environments as possible: sports environment, living environment, and disturbed environment. The exercise experiment was 3 times a week with a period of 12 weeks. The length of time was 40 minutes each time and a total experiment time of 1420 minutes. The music experiment was 3 times a week with a period of 12 weeks. The length of time was 40 minutes each time, and a total experiment time of 1420 minutes. Examples of songs：Everytime We Touch- Cascada (115 bpm), Beat It - Michael Jackson (120 bpm), Viva La
  Arms: experimental group of combine of exercise and music

SUMMARY:
The basic information collected in this study is based on demographic variables, including information such as class, gender, and age. In order to ensure the uniqueness of the participants and the consistency of the data before, during, and after the questionnaire, this study used the last six digits of the participant's student IDs for data collection. During the data collection phase, there was no phenomenon of the last six digits of the student ID being the same. This method ensured the correlation between the data before, during, and after the experiment, while protecting the privacy of the participants.

1. Experiment procedure In phase 2, this study recruited a total of 238 college students who volunteered to participate in this study. After screening according to the exclusion criteria, this study selected 108 eligible participants. This study included these 108 participants in the experiment of this study and randomly divided them into two groups, one for the experimental group and the other for the control group. In order to facilitate communication between the two groups of participants, this study created two WeChat groups, one for the experimental group and the other for the control group.

1.1 Experimental group: This study held a group meeting before the formal experiment to guide all participants in advance and describe the entire experimental process in detail to them. Students who had questions were given a unified and detailed explanation. Each participant received an instruction manual and a sports smart bracelet. During the experimental stage, the researcher would remind the participants on time to conduct the music and jogging experiment. The participants were required to participate in the experiment according to the contents of the instruction manual and upload each experimental participation content in the form of video or photos to the online information collection link posted by the participants. before experiment, 4 weeks, 8 weeks and 12 weeks，this study required participants to fill out the questionnaire four times.

1.2 Control group: At the same time as the experimental group, a booklet about music and exercise was distributed to the participants. The control group and the experimental group had the same time to fill in the questionnaire. The control group was asked to fill in the first questionnaire before the experiment. After 4 weeks, the control group was asked to fill in the second questionnaire. After 8 weeks, the control group was asked to fill in the third questionnaire. After 12 weeks, the control group was asked to fill in the fourth questionnaire。After the study completed, the control group was also provided with the music and jogging materials for their reference. So that they received the same benefit as the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. College students aged 18-24 years old;
2. Male and female,
3. Be in good health and free from major illness, measured by Physical Activity Readiness Questionnaire (PAR-Q).;
4. The group of Chinese college students' sports anxiety was screened according to the Chinese version of Physical Education and Sport Anxiety State (PESAS).

Exclusion Criteria:

1. College students who are not of Chinese nationality.
2. College students who are unwilling to participate in the experiment phase. College students who have any sports-related injuries.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Severity of exercise beliefs as Measured by the Exercise Beliefs Questionnaire | 12 weeks
  The Exercise Beliefs Questionnaire (EBQ) score for exercise beliefs. Possible scores range from 0 to 105, with higher scores indicating greater exercise beliefs.
Severity of sports anxiety as Measured by the Physical Education Sport Anxiety State Scale | 12 weeks
  The Physical Education Sport Anxiety State (PESAS) score for sports anxiety. Possible scores range from 0 to 90, with higher scores indicating a worse severity of sports anxiety.
Severity of mental toughness as Measured by the Mental Toughness For Youth Questionnaire | 12 weeks
  The Mental Toughness For Youth Questionnaire (MTYQ) score for mental toughness. Possible scores range from 0 to 175, with higher scores indicating greater mental toughness.
Severity of coping effectiveness as Measured by the Physical Education Sport Anxiety State Scale | 12 weeks
  The Coping Effectiveness (CE) score for coping effectiveness. Possible scores range from 0 to 35, with higher scores indicating greater coping effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Tourism College, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No